CLINICAL TRIAL: NCT00142454
Title: NY-ESO-1 Protein Vaccination in Malignant Melanoma Administered With Imiquimod as Adjuvant
Brief Title: NY-ESO-1 Protein Vaccine With Imiquimod in Melanoma (Adjuvant Setting)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2004-006; NYU 04-53 (Other: New York University)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Malignant Melanoma
Keywords: Malignant melanoma; Stages IIB-III
MeSH Terms: conditions — Melanoma | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imiquimod + NY-ESO-1 (Experimental): Patients applied topical imiquimod followed by vaccination with intradermal injections of the NY-ESO-1 protein.
  Interventions: Drug: Imiquimod; Biological: NY-ESO-1 protein

INTERVENTIONS:
Drug: Imiquimod — Patients applied imiquimod cream at bedtime every day for 5 consecutive days (for the first 5 days of Cycles 1-3 and for the first 4 days of Cycle 4) at a dose of 250 mg as supplied in single-use packets to a 4 x 5 cm area of healthy skin, alternating among the extremities (upper inner arms and inner thighs) in each cycle. The cream was to be rubbed into the skin until it was no longer visible. Patients were encouraged to wash their hands before and after applying cream. The application site was not occluded. The next morning, 6 to 10 hours after initial application, the treated area was washed with mild soap and water to remove any residual cream.
  Other Names: Aldara
Biological: NY-ESO-1 protein — NY-ESO-1 protein was injected intradermally by a study physician or nurse at a dose of 100 μg into the imiquimod-pretreated area on Day 3 of each cycle for 4 consecutive 21-day cycles.

SUMMARY:
This was a Phase 1, single-arm, open-label, pilot study of NY-ESO-1 protein vaccination with imiquimod as an adjuvant in patients with resected Stage IIB, IIC, and III malignant melanoma. The primary study objective was to determine the safety of NY-ESO-1 protein/imiquimod treatment, and the secondary objective was to evaluate the immunogenicity of treatment.

DETAILED DESCRIPTION:
Patients applied imiquimod (250 mg) topically to a designated area of healthy skin on the upper inner arm or inner thigh (the cream remained on the skin overnight for 6-10 hours) every day for 5 consecutive days (i.e., for the first 5 days of Cycles 1-3 and for the first 4 days of Cycle 4). The NY-ESO-1 protein (100 μg) was injected intradermally into the imiquimod-pretreated area on Day 3 of each cycle for 4 consecutive 21-day cycles.

Safety was monitored continuously. Immunization was assessed by the generation of NY-ESO-1-specific cluster of differentiation (CD)4+ and CD8+ T cell responses in enzyme-linked immunosorbent spot (ELISPOT) assays and by the development or augmentation of NY-ESO-1-specific antibody titers, assessed by enzyme-linked immunosorbent assay (ELISA).

Blood samples were obtained for the assessment of clinical biochemistry and hematology, and physical examinations were performed at baseline, on Day 1 of each cycle, and at a follow-up visit at Week 13.

Skin biopsies of the vaccinated area were obtained 48 hours after the last injection (Day 5 of Cycle 4). To avoid irritation, imiquimod was not applied after the biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Had histologically confirmed, resected American Joint Committee on Cancer Stage IIB, IIC or III malignant melanoma
* Fully recovered from surgery
* Age ≥ 18 years; children were excluded from this study, as the safety of imiquimod had not been established in patients below the age of 18
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate organ and marrow function as defined below:

  * absolute neutrophil count: ≥ 1500/μL
  * hemoglobin: ≥ 9 g/dL
  * platelets: ≥ 100,000/μL
  * total bilirubin: ≤ 1.5 × institutional upper limit of normal (ULN)
  * aspartate aminotransferase/alanine aminotransferase (AST/ALT): ≤ 2.5 × institutional ULN
  * creatinine: ≤ 1.5 × institutional ULN
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Received chemotherapy, immunotherapy (including interferon), or radiotherapy within 4 weeks prior to first dosing of study agent
* Prior treatment with NY-ESO-1 vaccines
* Known human immunodeficiency virus infection or autoimmune disease (rheumatoid arthritis, systemic lupus erythematosus), as these conditions could have interfered with the evaluation of the induced immune response; patients with vitiligo or melanoma-associated hypopigmentation were not excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to imiquimod or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection,symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would have limited compliance with study requirements
* Pregnancy or lactation
* Women of childbearing potential not using a medically acceptable means of contraception
* Known history of inflammatory skin disorders, as imiquimod might have exacerbated these conditions
* Chronic corticosteroid or immunosuppressive therapies, as these might have interfered with the evaluation of the induced immune response
* Lack of availability for immunological and clinical follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-08-24 (Actual); Primary Completion 2006-04-25 (Actual); Study Completion 2006-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD, PhD, Principal Investigator — NYU Langone Health; Sylvia Adams, MD, Study Director — NYU Langone Health
Locations (1):
- NYU Cancer Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adams S, O'Neill DW, Nonaka D, Hardin E, Chiriboga L, Siu K, Cruz CM, Angiulli A, Angiulli F, Ritter E, Holman RM, Shapiro RL, Berman RS, Berner N, Shao Y, Manches O, Pan L, Venhaus RR, Hoffman EW, Jungbluth A, Gnjatic S, Old L, Pavlick AC, Bhardwaj N. Immunization of malignant melanoma patients with full-length NY-ESO-1 protein using TLR7 agonist imiquimod as vaccine adjuvant. J Immunol. 2008 Jul 1;181(1):776-84. doi: 10.4049/jimmunol.181.1.776. PMID 18566444

RESULTS

PARTICIPANT FLOW:
Groups:
- Imiquimod + NY-ESO-1: Patients applied topical imiquimod cream (250 mg) to a designated area of healthy skin on the upper inner arm or inner thigh (the cream remained on the skin overnight for 6-10 hours) every day for 5 consecutive days (i.e., for the first 5 days of Cycles 1-3 and for the first 4 days of Cycle 4). A vaccination with the NY-ESO-1 protein (100 μg) was injected intradermally into the imiquimod-pretreated area on Day 3 of each cycle for 4 consecutive 21-day cycles.
Period: Overall Study
Arm/Group | Imiquimod + NY-ESO-1
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The population comprises all enrolled patients.
Arm/Group | Imiquimod + NY-ESO-1
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 49 [36 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 [Count of Participants; unit: Participants] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  Participants | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-emergent Adverse Events (TEAEs)
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0, as follows: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening), and Grade 5 (fatal). Adverse events (AEs) were reported based on clinical laboratory tests, vital sign and weight measurements, physical examinations, performance status evaluations, and any other medically indicated assessments, including patient interviews, from the time informed consent was signed through the last follow-up visit. AEs were considered to be treatment emergent (TEAE) if they occurred or worsened in severity after the first dose of study treatment.
Time Frame: Up to 4 months
Population: The population comprises all patients who received any dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Imiquimod + NY-ESO-1
Number analyzed (Participants) | 9
Participants
  Any TEAE | 8
  Maximum TEAE severity Grade 1 | 8
  Serious TEAE | 0
  TEAE leading to discontinuation | 0

2. Secondary Outcome: Number of Patients With Cellular Antibody Response to NY-ESO-1 at Two or More Post-vaccination Time Points
Description: Assays to assess cluster of differentiation (CD)8+ and CD4+ antigen-specific responses were performed at baseline (Cycle 1 Day 1), throughout the vaccination period (Day 1 of Cycles 2 through 4 and Day 10 of each cycle), and at the 2 post-treatment follow-up visits (Weeks 13 and 16) by enzyme-linked immune absorbent spot (ELISPOT) assay following prior in vitro sensitization. A 3-fold increase in spot-forming cells over baseline defined a positive response. Suitable antigens may have included recombinant viral vectors encoding NY-ESO-1, or NY-ESO-1 overlapping peptides, depending upon availability.
Time Frame: Up to 4 months
Population: The population comprises all patients who received any dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Imiquimod + NY-ESO-1
Number analyzed (Participants) | 9
Participants
  CD4+ T cell response | 7
  CD8+ T cell response | 0

3. Secondary Outcome: Number of Patients With Humoral Antibody Response to NY-ESO-1
Description: Assays to assess NY-ESO-1 specific antibodies were performed at baseline (Cycle 1 Day 1), throughout the vaccination period (Day 1 of Cycles 2 through 4 and Day 10 of each cycle), and at the 2 post-treatment follow-up visits (Weeks 13 and 16) by enzyme-linked immunosorbent assay (ELISA). Samples were diluted serially. The induction and augmentation of immunity were defined as an increase in antibody titer of ≥ 3× over buffer alone or ≥ 4× the pre-vaccination titer, respectively. Sera from the responding patients were tested a second time against a pool of NY-ESO-1 overlapping peptides to confirm NY-ESO-1 specificity; the number of patients in the table reflect the patients with confirmed NY-ESO-1 specificity.
Time Frame: Up to 4 months
Population: The population comprises all patients who received any dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Imiquimod + NY-ESO-1
Number analyzed (Participants) | 9
Participants | 4

ADVERSE EVENTS:
Time Frame: All adverse events (AEs), regardless of causality to study drug, were documented from informed consent through the final follow-up visit, which was up to 4 months for each patient.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 3.0), frequency, seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, preferred terms were counted only once per patient at the maximum reported grade.
Arm/Group | Imiquimod + NY-ESO-1
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 8/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imiquimod + NY-ESO-1 (N=9)
Redness at injection site (General disorders) | 6
Swelling at injection site (General disorders) | 2
Pain at injection site (General disorders) | 1
Splotchy at injection site (General disorders) | 1
Edema (General disorders) | 1
Boils (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Irregular heart rate (Cardiac disorders) | 1
Staph infection (Infections and infestations) | 1
Fatigue (General disorders) | 4
Tenderness on heel (General disorders) | 1
Itching at injection site (General disorders) | 1
Burning in groin area (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Hardness at injection site (General disorders) | 1
Flu-like symptoms (General disorders) | 2
Respiration infection (Infections and infestations) | 1
Injection site reaction (General disorders) | 2
Difficulty sleeping (Psychiatric disorders) | 1
Thigh pimple (Skin and subcutaneous tissue disorders) | 1
Mouth sores (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Itching shoulder scar (Skin and subcutaneous tissue disorders) | 1
Redness on thigh (Skin and subcutaneous tissue disorders) | 1
Flu shot reaction (General disorders) | 1
Redness on arm (Skin and subcutaneous tissue disorders) | 1
Leg edema (General disorders) | 1
Fever (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less